CLINICAL TRIAL: NCT00376038
Title: A Randomized Open-label, Repeat Dose, Two Sequence Cross-Over Study to Determine the Effect of GSK189075 on the Pharmacokinetic Parameters of Metformin (Glucophage) in Subjects With Type 2 Diabetes Mellitus.
Brief Title: Drug Interactions From Simultaneous Administration Of Metformin And GSK189075 To Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KG2105246
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: GSK189074; T2DM; GSK189075; Glucophage; Obesity; Diabetes; Metformin; Type 2 Diabetes Mellitus; Drug Interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Metformin

INTERVENTIONS:
Drug: GSK189075 oral tablets
Drug: metformin tablets
  Other Names: GSK189075 oral tablets

SUMMARY:
GSK189075 is intended for use as a single treatment or in combination with other treatments for tye 2 diabetes mellitus (T2DM). Metformin is widely used in Europe and the USA for the treatment of T2DM. This study will evaluate the effect of GSK189075 on metformin levels in the blood in T2DM subjects. The rationale is to look for any safety problems that may result when the 2 drugs are given together.

ELIGIBILITY:
Inclusion criteria:

* Have Type 2 diabetes mellitus.
* Have a Body Mass Index within range 22 to 35kg/m2 inclusive.
* Females who meet above criteria must be physiologically incapable of becoming pregnant (i.e., surgically sterilized, or post-menopausal per protocol definition).

Exclusion criteria:

* Are currently taking insulin therapy.
* Have any disease (such as heart, liver, blood, nervous system, or kidney disease, or cancer).
* Have a history of stomach, liver, kidney, or other disease that with interfere with taking the study drug.
* Are currently using diuretics, oral or injectable corticosteroids (inhaled & intranasal corticosteroids are permitted), or other medications that would cause you to deplete your fluid balance in your body; currently taking stable regimens for heart conditions; currently using prescription or non-prescription drugs within 7 days of starting the study that may interfere with the study drug.
* Would donate more than 450 ML of blood over a 2 month period.
* Physician does not think it is a good idea for you to participate in the trial. - Had a urinary tract infection or bladder infection in the last month. - Are currently drinking more than 2 beers, 1 glass of wine, or 1 glass of spirits daily.
* Have a positive urine drug screen test.
* Plan to change your smoking habits during the course of the trial.
* Have Hepatitis C, Hepatitis B, or HIV. - Have a lab or EKG abnormality. - High or low blood pressure.
* Have used of any investigational drug or device during the study or within 30 days prior to 1st dosing of study medication.
* Are a male subject unwilling to abstain or use protection during intercourse.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Blood concentrations of metformin when given with GSK189075 in T2DM subjects over 3-day course Lab tests, changes in blood pressure and heart rate and heart activity on EKG machine

SECONDARY OUTCOMES:
Blood levels of drugs at Day 3 Evaluation of efficacy and safety markers on Days 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mexico City, Mexico

REFERENCES:
- [Derived] Hussey EK, Kapur A, O'Connor-Semmes R, Tao W, Rafferty B, Polli JW, James CD Jr, Dobbins RL. Safety, pharmacokinetics and pharmacodynamics of remogliflozin etabonate, a novel SGLT2 inhibitor, and metformin when co-administered in subjects with type 2 diabetes mellitus. BMC Pharmacol Toxicol. 2013 Apr 30;14:25. doi: 10.1186/2050-6511-14-25. PMID 23631443